CLINICAL TRIAL: NCT00963768
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Oral Doses of JNJ-28431754 in Type 2 Diabetes Mellitus Patients
Brief Title: A Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of JNJ-28431754 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR012451; 28431754NAP1002 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; JNJ-28431754; Canagliflozin; Sodium Glucose Co-transporter (SGLT2 inhibitor); Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): JNJ-28431754 30 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: JNJ 28431754; Drug: Placebo
- Cohort 2 (Experimental): JNJ-28431754 100 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: JNJ 28431754; Drug: Placebo
- Cohort 3 (Experimental): JNJ-28431754 300 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: JNJ 28431754; Drug: Placebo
- Cohort 4 (Experimental): JNJ-28431754 600 mg/day or placebo. The actual dose (mg) level selected for each cohort may be modified based on evaluation of preliminary safety, pharmacokinetic and pharmacodynamic data from previous cohorts.
  Interventions: Drug: JNJ 28431754; Drug: Placebo
- Cohort 5 (Experimental): JNJ-28431754 at 30 mg/day, 100 mg/day, or 300 mg/day or placebo (the dose level to be determined from the prior cohort of patients tested and considered to be well tolerated).
  Interventions: Drug: JNJ 28431754; Drug: Placebo

INTERVENTIONS:
Drug: JNJ 28431754 — A liquid suspension of 30 mg, 100 mg, 300 mg of JNJ-28431754 taken once (or twice) daily or 600 mg taken once daily will be administered by study personnel directly into the patient's mouth using an oral liquid dispenser for 14 days (Day 1 and Days 3 through 16).
  Other Names: Canagliflozin
Drug: Placebo — A liquid suspension of placebo will be administered by study personnel directly into the patient's mouth using an oral liquid dispenser once or twice daily for 14 days (Day 1 and Days 3 through 16).

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (ie, blood levels of JNJ-28431754) and pharmacodynamics (ie, urine and blood levels of glucose) of JNJ-28431754 compared to placebo in patients with Type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither physician, patient nor the sponsor knows the assigned treatment), placebo-controlled, single and multiple (14 days) ascending dose, parallel group study in 3 study centers (United States, Germany and South Korea). Five cohorts (groups) of patients with Type 2 diabetes mellitus (T2DM) will be studied. One dose level will be evaluated in each cohort. Sixteen (16) patients will be randomly assigned to receive JNJ-28431754 and four (4) patients to receive matching placebo within each cohort. The planned doses are 30, 100, 300 and 600 mg per day. Twice-daily dosing may also be evaluated in one or more of the cohorts. An additional cohort of Asian patients will also be evaluated at a dose level, which was previously tested in a prior cohort and considered to be well tolerated. Blood and urine samples will be collected from patients during the study for pharmacokinetic and pharmacodynamic assessments. The safety and tolerability of JNJ-28431754 will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with Type 2 Diabetes for at least one year before screening
* Patients must be taking a stable dose of oral (by mouth) anti-diabetic monotherapy or a combination of two anti-diabetic medications
* Males or postmenopausal or surgically sterile women (post-menopausal is defined as no menses for at least 18 months prior to study start or no menses for 6 to 18 months)
* Body mass index (weight in kg/height in m2) should be between 20 to 39.9 kg/m2

Exclusion Criteria:

* History of Type 1, brittle diabetes or secondary forms of diabetes
* History of repeated severe hypoglycemic episodes
* History of diabetic complications including retinopathy, nephropathy, neuropathy, gastroparesis, or ketoacidosis
* History of, or currently active illness including but not limited to cardiovascular disease, hematological disease, respiratory disease, hepatic or gastrointestinal disease, endocrine/metabolic disorders, neurologic or psychiatric disease, or malignant neoplasms considered by the Investigator to be clinically significant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The number of patients with adverse events as a measure of safety and tolerability | Up to 34 days (baseline [Day -1] through follow up [10 days following Day 22 visit])

SECONDARY OUTCOMES:
Change from baseline (Day -1) for mean 24-hour plasma glucose concentration | Day -1 through Day 16
Change from baseline 24-hour urinary glucose excretion (UGE) | Day -1 through 16
Change from baseline mean fasting plasma glucose | Day -1 through Day 16
Change from baseline mean morning fasting body weight | Day -1 through 20
Renal glucose threshold | Day -1 through Day 16

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (3):
- Chula Vista, California, United States
- Neuss, Germany
- Seoul, South Korea

REFERENCES:
- [Derived] Sha S, Devineni D, Ghosh A, Polidori D, Hompesch M, Arnolds S, Morrow L, Spitzer H, Demarest K, Rothenberg P. Pharmacodynamic effects of canagliflozin, a sodium glucose co-transporter 2 inhibitor, from a randomized study in patients with type 2 diabetes. PLoS One. 2014 Sep 30;9(9):e110069. doi: 10.1371/journal.pone.0110069. eCollection 2014. PMID 25268802
- [Derived] Sha S, Devineni D, Ghosh A, Polidori D, Hompesch M, Arnolds S, Morrow L, Spitzer H, Demarest K, Rothenberg P. Pharmacodynamic effects of canagliflozin, a sodium glucose co-transporter 2 inhibitor, from a randomized study in patients with type 2 diabetes. PLoS One. 2014 Aug 28;9(8):e105638. doi: 10.1371/journal.pone.0105638. eCollection 2014. PMID 25166023
- See also: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Oral Doses of JNJ-28431754 in Type 2 Diabetes Mellitus Patients — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=747&filename=CR012451_CSR.pdf